CLINICAL TRIAL: NCT00161837
Title: Single-blind Randomized Controlled Phase II/III Study to Investigate the Immunogenicity and Safety of an Inactivated Influenza Vaccine (Whole Virion, Vero Cell Derived) in Comparison to a Licensed Egg-derived Influenza Vaccine for Season 2003/2004
Brief Title: Comparison of the Safety and Immune Response of an Influenza Vaccine Made by a New Manufacturing Process With a Vaccine Made by the Traditional Manufacturing Process for Season 2003/2004
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 227
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2006-10

CONDITIONS: Influenza
Keywords: Influenza; Vaccine
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Vero Cell-derived Influenza Vaccine
Biological: Egg-derived Influenza Vaccine

SUMMARY:
The objectives of the study are to assess the immunogenicity and safety of the inactivated influenza vaccine (whole virion, Vero cell-derived) at Day 21 and Day 180 after vaccination.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects will be eligible for participation in this study if they:

* are >= 18 and <= 60 years old (for Stratum A only);
* are > 60 years old (for Stratum B only);
* are in a physical condition such that the physician would have no reservations vaccinating with an influenza vaccine outside the scope of a clinical trial;
* will reliably keep a daily record of symptoms;
* understand the nature of the study, agree to its provisions, and give written informed consent;
* if female and capable of bearing children - show a negative pregnancy test result at study entry and agree to employ adequate birth control measures for the duration of the study.

Exclusion Criteria:

Male and female subjects will be excluded from participation in this study if they:

* have received any influenza vaccine for the 2002/2003 season and/or for the 2003/2004 season;
* suffer from any kind of immunodeficiency;
* suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids, chemotherapeutics) that can be expected to influence immunological functions;
* have a history of inflammatory or degenerative neurological disease (e.g. Guillain Barré, multiple sclerosis);
* have received a blood transfusion or immunoglobulins within one month of study entry;
* have a history of any vaccine-related contraindicating event (e.g. anaphylaxis);
* have a rash or dermatological condition which may interfere with injection site reaction rating;
* have a known or suspected problem with drug or alcohol abuse;
* are unable to lead an independent life either physically or mentally;
* had administration of an investigational drug within six weeks prior to the study start;
* are concurrently participating in a clinical trial;
* are pregnant or lactating.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-12; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Romaszko, MD, Principal Investigator — PANTAMED sp. z o o.
Locations (1):
- PANTAMED Sp.z o.o., Olsztyn, Poland